CLINICAL TRIAL: NCT05069701
Title: The Effect of Different Head and Trunk Positions on Static Virtual SVV and Dynamic Virtual SVV in Healthy Individuals: A Standardization Study
Brief Title: The Effect of Different Head and Trunk Positions on SVV in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Fazıl Necdet Ardıç, Professor, Pamukkale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9
Record Dates: First submitted 2021-09-26; First posted 2021-10-06 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-01

CONDITIONS: Virtual Reality

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteers (Experimental): SVV test will be done.
  Interventions: Diagnostic Test: SVV test

INTERVENTIONS:
Diagnostic Test: SVV test — SVV test will be done with virtual reality glasses.

SUMMARY:
Aim: To obtain standardization data in static virtual SVV and dynamic virtual SVV tests according to different head and body positions by keeping up with developing technologies. In this way, it is planned to evaluate the treatment responses of patients who receive vestibular rehabilitation in a healthier way.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult volunteers
2. Volunteers over 18 years old

Exclusion Criteria:

1. Patients with impaired cooperation
2. Musculoskeletal or systemic presence of disease
3. Past ear disease
4. Patients who have experienced dizziness
5. Presence of central nervous system pathology
6. Patients who have used ototoxic drugs
7. Patients whose use of glasses may cause problems (epilepsy, vision loss, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-07-10 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
Static SVV test | 1 month
  For commercially available VR Subjective Visual vertical(SVV), VIRTUALIS® PHYSIO VR[SVV and Dynamic SVV](Virtualis, France) was used. The bar angles are given in a random order. The system consists of glasses, computer and hand control. When patients wear their glasses, they can see only a light bar in Static SVV, and points rotating left or right on the background of the light bar in Dynamic SVV. No light can enter the glasses. The glasses have a sensor that detects the angle of the head. The starting point of the bar can be adjusted randomly to different angles by the computer. The visual background rotation rate for dynamic SVV was determined as ±30°/sec. The subject should adjust the bar in the vertical position using the right/left arrows on the controller. When verticality is confirmed by pressing the set button in the middle of the control unit, the computer records the angle of the bar and the position of the head.
Dynamic SVV test | 1 month
  For commercially available VR Subjective Visual vertical(SVV), VIRTUALIS® PHYSIO VR[SVV and Dynamic SVV](Virtualis, France) was used. The bar angles are given in a random order. The system consists of glasses, computer and hand control. When patients wear their glasses, they can see only a light bar in Static SVV, and points rotating left or right on the background of the light bar in Dynamic SVV. No light can enter the glasses. The glasses have a sensor that detects the angle of the head. The starting point of the bar can be adjusted randomly to different angles by the computer. The visual background rotation rate for dynamic SVV was determined as ±30°/sec. The subject should adjust the bar in the vertical position using the right/left arrows on the controller. When verticality is confirmed by pressing the set button in the middle of the control unit, the computer records the angle of the bar and the position of the head.

CONTACTS AND LOCATIONS:
Overall Officials: Fazıl Necdet Ardıç, Professor, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)